CLINICAL TRIAL: NCT01275443
Title: A Pharmacokinetic Evaluation of the Exposure and Distribution of TMC278LA for Use as Pre-exposure Prophylaxis, in Plasma and Genital Tract / Rectal Compartments, Following a Single Intramuscular Dose at Different Doses in HIV-negative Healthy Volunteers.
Brief Title: Study in Healthy Volunteers of the Safety and Metabolism of Different Doses of the Anti-HIV Drug TMC278LA.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SSAT 040
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: HIV Infection
Keywords: HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 300mg TMC278LA (Experimental): Single gluteal intramuscular injection (300mg) at day 1
  Interventions: Drug: 300mg TMC278LA
- 1200mg TMC278LA (Experimental): Single gluteal intramuscular injection (1200mg) at day 1
  Interventions: Drug: 1200mg TMC278LA
- 600mg TMC278LA (Experimental): Single gluteal intramuscular injection (600mg) at day 1
  Interventions: Drug: 600mg TMC278LA
- 150mg TMC278LA (Experimental): This arm was included in the adaptive design of the study, but was not recommended for use based on the review of results from 300mg and 600mg arms by the protocol steering committee
  Interventions: Drug: 150mg TMC278LA

INTERVENTIONS:
Drug: 300mg TMC278LA — 300mg TMC278LA intramuscular injection
  Other Names: rilpivirine long-acting
  Arms: 300mg TMC278LA
Drug: 150mg TMC278LA — 150mg TMC278LA intramuscular injection
  Other Names: rilpivirine long-acting
  Arms: 150mg TMC278LA
Drug: 1200mg TMC278LA — 1200mg TMC278LA intramuscular injection
  Other Names: rilpivirine long-acting
  Arms: 1200mg TMC278LA
Drug: 600mg TMC278LA — 600mg TMC278LA intramuscular injection
  Other Names: rilpivirine long-acting
  Arms: 600mg TMC278LA

SUMMARY:
TMC278 (also called rilpivirine) is a new drug being developed to treat HIV. Usually TMC278 is taken as a tablet, by mouth, once a day, but a 'long acting' formulation has been developed so the drug stays in the bloodstream for a longer time - this allows the drug to be given by injection and less often. It is hoped that this injectable version of the drug may be used to help prevent HIV transmission in the future by giving it to people who are at risk of HIV. This is similar to the way travellers to areas with malaria may take antibiotics to prevent infection. The investigators aim to investigate the feasibility of using TMC278 as a preventative medication by performing this study.

The purpose of this study is to investigate the levels of drug which can be measured in the blood, as well as the tissues and fluids of the rectum (the lowest part of the bowels just before the opening of the anus) as well as the safety of the drug and how well tolerated it is when given as a single dose. In this study, the investigators will not be investigating whether the drug prevents HIV so the investigators will recruit people who are HIV negative, and whose lifestyle does not put them at risk of becoming infected before or during the study.

If the study shows the drug is well tolerated and produces appropriate levels of the drug (in the bloodstream and the rectal compartment) to suggest that it could be effective, it will help design future studies looking at preventing HIV.

DETAILED DESCRIPTION:
The trial will examine the pharmacokinetics of doses of 300mg and 600mg, as well as either 150mg or 1200mg, of TMC278LA, given as a single intramuscular dose to HIV-negative participants. Investigation of drug pharmacokinetics in plasma, female genital secretions and tissue samples, and male rectal fluid and tissue samples (at the 600mg dose) will be also carried out in order to provide data on relative drug exposure following drug administration. Additionally, ex-vivo assays to assess viral inhibition in fluid from genital secretions and rectal compartments will provide partial information on pharmacodynamic characteristics of TMC278; this may usefully inform future selection decisions on the appropriate target concentrations required for prevention.

The target concentration for a prophylactic use of TMC278 in plasma, genital or rectal tissues and fluids is unknown. It is possible that a target lower than that required for treatment of established infection would be suitable. However, there is currently no pharmacodynamic data to usefully inform what this target concentration might be. In the absence of population PK data in an efficacy trial of TMC278 as a prophylactic agent, the investigators aim to obtain useful indirect data from ex-vivo viral inhibition assays to at least guide future decisions on dose selection.

Up to 60 evaluable female participants will be enrolled, with more than 40% being of African ancestry. Six male participants will also be enrolled. This will provide data on plasma pharmacokinetics and the relative distribution kinetics in the female genital tract and male rectal compartment in order to support expanded safety studies and a phase III global efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

1. The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all trial requirements.
2. Non-pregnant, non-lactating females (at least 40% will be of self-identified African ancestry)
3. Age between 18 to 50 years, inclusive.
4. Body Mass Index (BMI) of 16 to 35 kg/m2, inclusive.
5. Negative antibody/antigen combined test for HIV1 and HIV2.
6. Absence of any significant health problems (in the opinion of the investigator) on the basis of the screening procedures; including medical history, physical examination, vital signs, ECG.
7. Willing to undergo HIV testing, HIV discussion and receive HIV test results throughout the trial (according to the "UK National Guidelines for HIV Testing 2008", www.bhiva.org).
8. Women of childbearing potential (WOCBP) must be using an adequate method of contraception (intrauterine device, condoms, anatomical sterility in self or partner) to avoid pregnancy throughout the trial and for a period of at least four months after the trial follow up visit (oral hormonal methods and implant contraceptives are allowed but only in combination with the additional protection of a barrier method). Males participating in sexual intercourse that could result in pregnancy must use condoms during the duration of the study and for up to four months following the follow up visit.
9. Willing to abstain from sexual intercourse (vaginal for females and receptive anal for males) for 48 hours prior to each trial visit (with complete abstinence in the first 28 days post-dose).
10. Females willing to refrain from the use of vaginal products or objects including, tampons, female condoms, cotton wool, rags, diaphragms, cervical caps (or any other vaginal barrier method), douches, lubricants, vibrators/dildos, and drying agents for 14 days prior to enrolment and for the duration of the trial. Males willing to refrain from the use of anal products or objects including douches, lubricants and vibrators/dildos for 14 days prior to enrolment and for the duration of the trial.
11. Likely to remain resident in the UK for the duration of the trial period.
12. Willing to consent to their personal details being entered onto The Over volunteering Prevention Scheme (TOPS) database.
13. Willing to provide photographic identification at each visit.
14. Registered with a GP in the UK

Exclusion Criteria:

1. Any significant acute or chronic medical illness.
2. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations.
3. Positive blood screen for syphilis, hepatitis A (IgM) B (HBs Ag) and/or C antibodies.
4. Positive blood screen for HIV-1 and/or HIV-2 antibodies.
5. Positive screen for sexually transmitted infections at screening visit (if bacterial vaginosis or candidiasis detected at screen, these may be treated with test-of-cure prior to enrolment).
6. Prolonged QT interval on screening ECG, or clinically significant change as judged by investigator.
7. High-risk behaviour for HIV infection which is defined as having one of the following within six months before trial day 0 (first dose):

   i. had unprotected vaginal or anal sex with a known HIV infected person or a casual partner.

   ii. engaged in sex work for money or drugs. iii. acquired a sexually transmitted disease. iv. having a high risk partner either currently or in the previous six months
8. Clinically relevant alcohol or drug use (positive urine drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events.
9. Exposure to any investigational drug or placebo within 30 days of first dose of trial drug (additional check to be made on TOPS www.tops.org.uk).
10. History of severe drug allergy that in the opinion of the Investigator may increase the risk of developing an allergic reaction to the trial drug.
11. Use of any drug, including over-the-counter medications and herbal preparations, within two weeks prior to first dose of trial drug (unless approved or prescribed by the Investigator (for exceptions see section 5.2).
12. Females who are pregnant or breast-feeding..
13. Clinically significant laboratory abnormalities (according to normal range as defined by central laboratory).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetics | 84 days
  The plasma pharmacokinetics of TMC278LA at different dose levels up to 84 days after a single intramuscular administration
TMC278LA concentrations in the genital tract and rectal compartments. | 84 days
  TMC278LA concentrations in the genital tract and rectal compartments following the administration of different doses in HIV-negative healthy volunteers.

SECONDARY OUTCOMES:
Safety and tolerability of TMC278LA | 84 days
  The safety and tolerability of up to four different doses of TMC278LA administered as a single dose intramuscularly assessed by clinical and laboratory tests and adverse event reporting
HIV replication in vitro | 84 days
  The effect of the genital and rectal fluid drug concentrations on HIV replication in vitro (pharmacodynamic [PD] analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Dr, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- St Stephen's AIDS Trust, London, United Kingdom

REFERENCES:
- [Result] Jackson AG, Else LJ, Mesquita PM, Egan D, Back DJ, Karolia Z, Ringner-Nackter L, Higgs CJ, Herold BC, Gazzard BG, Boffito M. A compartmental pharmacokinetic evaluation of long-acting rilpivirine in HIV-negative volunteers for pre-exposure prophylaxis. Clin Pharmacol Ther. 2014 Sep;96(3):314-23. doi: 10.1038/clpt.2014.118. Epub 2014 May 26. PMID 24862215